CLINICAL TRIAL: NCT03660644
Title: Physical Activity Following Pulmonary Rehabilitation in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Physical Activity Following Pulmonary Rehabilitation in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Collaborators: National Health Service, United Kingdom (Other Government); British Lung Foundation (Other); University College, London (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 180203
Record Dates: First submitted 2018-05-17; First posted 2018-09-06 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-09

CONDITIONS: COPD; Physical Activity
Keywords: COPD; Physical Activity; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Physiotherapists will be aware of the allocation of the programmes (not possible to blind) as they will be involved with delivering information/training of the intervention components. However, a researcher blinded to group allocation will perform the quantitative analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WhatsApp, Pedometer and Step Diary (Experimental): Pedometer, step diary and WhatsApp following pulmonary rehabilitation
  Interventions: Behavioral: WhatsApp, Pedometer and Step Diary
- Control (No Intervention): Usual care following pulmonary rehabilitation.

INTERVENTIONS:
Behavioral: WhatsApp, Pedometer and Step Diary — Participants will be provided with a daily step diary and added to a group chat on WhatsApp. The group chat will be populated by other members of pulmonary rehabilitation programme (cluster) and the WhatsApp group leader will encourage participants to keep active. Participants will be encouraged to record the number of steps walked in a paper diary at the end of each day (i.e. prior to bedtime). This diary will simply have three columns: day of the week; number of steps; comments (optional).
  The intervention will last 52 weeks.
  Arms: WhatsApp, Pedometer and Step Diary

SUMMARY:
The aim of this feasibility study is to identify the acceptability of an intervention designed to promote physical activity following pulmonary rehabilitation for individuals with Chronic Obstructive Pulmonary Disease (COPD). Participants in the intervention group will be provided with pedometers and step diaries and added to a WhatsApp group with other graduates of pulmonary rehabilitation for 52 weeks.

DETAILED DESCRIPTION:
Evidence suggests that physical activity is not maintained following pulmonary rehabilitation for individuals with COPD. Peer social support, feedback about physical progression and recognition of opportunities to stay active following pulmonary rehabilitation have been identified as facilitators to physical activity following pulmonary rehabilitation. The proposed feasibility study has incorporated these factors into the intervention.

This is a mixed-methods study including a feasibility cluster randomised controlled trial and a qualitative process evaluation. Clusters will be pulmonary rehabilitation programmes across Lincolnshire Community Health Services, NHS Trust (n=8), randomly allocated to the Intervention or Control. Patients in the Intervention group will receive a multi component intervention following pulmonary rehabilitation (pedometer, step diary and WhatsApp) and patients in the Control group will receive standard care following pulmonary rehabilitation.

The primary objective is to identify and report the acceptability of the intervention for patients. The secondary objectives are to: 1) gather information on recruitment and consent rates of patients who are eligible and willing to participate, and to monitor retention of participants throughout the study; 2) understand the patients' and health care professionals' experience and views of the intervention and research procedures; 3) identify and report intervention fidelity throughout the study; 4) provide an estimate of likely changes in the proposed primary outcome for the full randomised controlled trial (average daily step count at 52 weeks following pulmonary rehabilitation) and other secondary health outcomes; 5) obtain the necessary statistical parameters to inform sample size calculations in a future definitive cluster randomised controlled trial. The results from the feasibility study will inform the design of a definitive trial, including whether the specific intervention has the potential to promote physical activity.

ELIGIBILITY:
Inclusion Criteria:

Cluster level

* Pulmonary rehabilitation programmes within Lincolnshire Community Health Services (NHS trust).
* Permission from the lead healthcare professionals of the pulmonary rehabilitation programme for the programme to be involved in the study.

Patient level

* Adults (age range: 30-100 years) with COPD who are enrolled in pulmonary rehabilitation within Lincolnshire Community Health Services (NHS trust).
* Provide informed consent for their outcome data to be collected.

Patients (for telephone interviews)

* Have access to a telephone.
* Adults (age range: 30-100 years) with COPD who are enrolled in pulmonary rehabilitation within Lincolnshire community health services (NHS trust).
* Provide informed consent to participate in a telephone interview (including patients who do/do not consent for their outcome data to be collected).

Health care professionals

* Involved in delivering the pulmonary rehabilitation programmes allocated to the Intervention Group within Lincolnshire Community Health Services (NHS trust).
* Provide informed consent to participate in a focus group.

WhatsApp group leaders

* Volunteers (who were members of local COPD support groups, whom held the position of Chair, Treasurer or Secretary, or were ordinary members, and in general, sufficiently stable to be a proactive and regular member of the group)
* Provide informed consent to lead the WhatsApp groups.

Exclusion Criteria:

Cluster level

* Pulmonary rehabilitation programmes which are not within Lincolnshire Community Health Services (NHS trust).
* The lead health care professionals of the pulmonary rehabilitation programmes are unwilling for the programme to be involved in the study.

Patient level

* Not enrolled on a pulmonary rehabilitation programme within Lincolnshire Community Health Services (NHS trust) or those who drop out of pulmonary rehabilitation following enrolment.
* Unable/unwilling to provide informed consent for their outcome data to be collected.
* Involved in another research study including the use of an intervention to promote physical activity.

Patients (telephone interviews)

* Do not have access to a telephone.
* Not enrolled on a pulmonary rehabilitation programme within Lincolnshire Community Health Services (NHS trust) or those who drop out of pulmonary rehabilitation following enrolment.
* Unable/unwilling to provide informed consent to participate in a telephone interview.

Health care professionals

* Not involved in delivering the pulmonary rehabilitation programmes allocated to the Intervention Group.
* Unable/unwilling to provide informed consent to participate in a focus group.

WhatsApp group leaders

* Not volunteers (and have not been involved in local COPD support groups, have not held the position of Chair, Treasurer or Secretary, have not been ordinary members, and in general, are not sufficiently stable to be a proactive and regular member of the group)
* Unable/unwilling to provide informed consent to lead the WhatsApp groups.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention | 55 weeks
  The number of patients who comply with the intervention will be measured

SECONDARY OUTCOMES:
Recruitment rates | Up to 26 weeks (approximately)
  The time taken to achieve planned sample size (clusters, participants) will be measured
Consent rates | Up to 26 weeks (approximately)
  The number of eligible patients willing to consent to take part in the study will be measured
Attrition rates | Up to 55 weeks (study completion)
  The number of patients who withdraw from the study will be measured
Semi-structured telephone interviews with subsets of patients | At relevant intervals up to 55 weeks (study completion)
  Patients' experience/views of the research procedures and intervention will be measured
Focus groups with health care professionals | At relevant intervals up to 55 weeks (study completion)
  Healthcare professionals' experience/views of the research procedures and intervention will be measured
Content of anonymised WhatsApp chat | At 4 week intervals, up to 55 weeks (study completion)
  The WhatsApp chats will be sent to the research team to measure intervention fidelity.
WhatsApp Checklist | At 4 week intervals, up to 55 weeks (study completion)
  The WhatsApp checklists will be sent to the research team to measure the intervention fidelity.
Step diary (self-reported) | 55 weeks (study completion)
  Patients' step diaries will be collected to assess the intervention fidelity.
Activity levels | During pulmonary rehabilitation (baseline), 12 and 52 weeks after pulmonary rehabilitation
  Activity levels will be measured by an activity monitor (Actigraph wGT3X-BT). Physical activity will be specified for:
  1. Time spent in different activity intensities
  2. Time spent sedentary
  3. Daily and weekly steps
  4. Weekly Vector Magnitude Units
PROactive tool | During pulmonary rehabilitation (baseline); 12 and 52 weeks after pulmonary rehabilitation
  The PROactive tool measures both physical activity amount (from the activity monitor) and physical activity difficulty to compute a reliable measure of physical activity in COPD.
Sleep levels | Baseline, 12 and 52 weeks after pulmonary rehabilitation
  Sleep will be measured by an activity monitor (Actigraph wGT3X-BT).
  Sleep will be specified for:
  1. Sleep latency
  2. Total sleep time
  3. Wake after sleep onset
  4. Sleep efficiency.
Sleep (self-reported sleep habits) | During pulmonary rehabilitation (baseline), 12 and 52 weeks after pulmonary rehabilitation
  In conjunction with wearing an activity monitor, participants will report the:
  1. Time went to bed
  2. Time taken to fall asleep
  3. Time woke up
Incremental Shuttle Walk Test (ISWT) | During pulmonary rehabilitation (baseline), 12 and 52 weeks after pulmonary rehabilitation
  The ISWT will measure participants functional capacity.
Chronic Respiratory Questionnaire (CRQ) | During pulmonary rehabilitation (baseline); 12 and 52 weeks after pulmonary rehabilitation
  The CRQ will measure patients' disease specific quality of life.
Hospital Anxiety and Depression Scale (HADS) | During pulmonary rehabilitation (baseline); 12 and 52 weeks after pulmonary rehabilitation
  HADS will measure patients' psychological well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Robinson, MSc, Principal Investigator — University of Lincoln
Locations (1):
- NHS pulmonary rehabilitation clinics across Lincolnshire, Lincoln, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No